CLINICAL TRIAL: NCT06227806
Title: Surgery and Exercise Versus Exercise Only for Chronic Patellofemoral Pain Syndrome: a Randomised Controlled Trial
Brief Title: Surgery and Exercise Versus Exercise Only for Chronic Patellofemoral Pain Syndrome
Acronym: REVITALISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canisius-Wilhelmina Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL80956.091.22
Record Dates: First submitted 2024-01-09; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Patellofemoral Pain Syndrome; Tibial Tubercle Transfer; Home Exercise Program
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tibial Tubercle Transfer surgery (Experimental): Tibial Tubercle Transfer surgery followed by a home exercise program.
  Interventions: Procedure: Tibial Tubercle Transfer
- Home Exercise Program (Active Comparator): A home exercise program.
  Interventions: Procedure: Home Exercise Program

INTERVENTIONS:
Procedure: Tibial Tubercle Transfer — Patients will receive the TTT surgery followed by a home exercise program.
  Arms: Tibial Tubercle Transfer surgery
Procedure: Home Exercise Program — Patients will receive an extensive home exercise program.
  Arms: Home Exercise Program

SUMMARY:
The goal of this randomised controlled trial is to compare a tuberositas transposition (TTT) surgery with a home exercise program (HEP) in patients with patellofemoral pain syndrome (PFPS). The study aims to evaluate the efficiency of TTT in conjunction with a HEP compared to a HEP alone in patients with chronic PFPS.

Participants will randomly be allocated to the surgery or HEP group. Researchers will compare the surgery and HEP groups to see if activity-related pain and patient reported outcome measures (PROMs) are different.

ELIGIBILITY:
Inclusion Criteria:

* Characteristic history of PFPS (patellofemoral pain during knee loading physical activity, such as jumping, running, squatting);
* Symptoms lasting at least 12 months;
* Tibial tubercle trochlear groove (TT-TG) distance of 15mm or more on CT or MRI;
* Patellofemoral pain during daily life activities, such as: standing for an extended period, walking, or walking upstairs or downstairs

Exclusion Criteria:

* Previous knee surgery;
* Reported knee ligamentous or meniscal injuries;

  * Disabling general illness;
  * A history of patellar dislocation; however, subjects with patellar subluxation are included in the study;
  * Other knee problems than PFPS diagnosed clinically (such as jumper's knee);
  * Other knee problems than PFPS diagnosed radiographically (such as osteochondritis - dissecans);
  * Patients who cannot undergo surgery;
  * Pregnancy;
  * Patients with inability to complete follow-up or with limited understanding of the Dutch language

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue pain score (VAS) | baseline and 12 weeks after HEP or 18 weeks after TTT surgery
  10-cm (0-10) visual VAS to assess activity-related pain. Higher scores reflect higher pain.

SECONDARY OUTCOMES:
Kujala pain score | baseline, after 12 weeks after HEP or 18 weeks after TTT surgery, 26 weeks, and 1 year
  The Kujala Score or Anterior Knee Pain Scale (AKPS) is a 13-item questionnaire to evaluate subjective symptoms and functional limitations in patients with PFP. The AKPS is graded on a scale of 0-100, with 100 reflecting no signs of PFP.
International Knee Documentation Committee Subjective Knee Form (IKDC) | baseline, after 12 weeks after HEP or 18 weeks after TTT surgery, 26 weeks, and 1 year
  The IKDC is a tool containing 7 items on knee symptoms, 2 on function, and 2 on sports activities, resulting in a score from 0-100, with 100 reflecting the highest level of pain and functional restrictions.
Tegner Activity Score | baseline, after 12 weeks after HEP or 18 weeks after TTT surgery, 26 weeks, and 1 year
  The Tegner Activity Score consists of 1 item, scoring the level of work- and sport activities, which is scored by a 10-point scale with 10 reflecting high level of activity.
EuroQol health-related quality of life (EQ-5D-5L) questionnaire | baseline, after 12 weeks after HEP or 18 weeks after TTT surgery, 26 weeks, and 1 year
  The health-related quality of life (EQ-5D-5L) questionnaire consists of states of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that are scored on 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems). An index value will be calculated to reflect health state on a scale of 0 to 1, where 1 represents maximum quality of life.
Visual analogue pain score (VAS) | after 6 weeks, 26 weeks, and 1 year
  10-cm (0-10) visual VAS to assess activity-related pain. Higher scores reflect higher pain.
Knee functionality using Decline step down test (DSDT) | baseline and after 26 weeks
  The DSDT is a performance test simulating stair descent. It assesses maximum pain-free flexion angle, from 0 to 90 degrees. Larger angles reflect higher functionality of the knee.

CONTACTS AND LOCATIONS:
Overall Officials: Sander Koëter, PhD, Principal Investigator — Canisius-Wilhelmina Hospital
Locations (1):
- Canisius Wilhelmina Hospital, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The trial protocol is available from the corresponding author on reasonable request. Data will be handled according to the FAIR principles. After completion of the study, metadata will be available upon request. For access to participant level-data and statistical code, an application can be submitted to the corresponding author.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication of the results of the study in a scientific article, data will become available for 15 years.
Access Criteria: Reasonable request.

REFERENCES:
- [Derived] van de Ven MPF, Ophey M, van de Graaf V, van de Groes SAW, Sinkeldam M, Wijers CHW, Koeter S. Tibial tubercle transfer SurgeRy and physiothErapy Versus physIotherapy only for chronic paTellofemorAL paIn: study protocol for a randomiSed controllEd trial (REVITALISE). BMC Musculoskelet Disord. 2025 Jan 15;26(1):53. doi: 10.1186/s12891-024-08226-y. PMID 39815178